CLINICAL TRIAL: NCT00168974
Title: Somatosensoric and Autonomic Disturbances in Female Patients With Fabry Disease
Brief Title: Neuropathic Pain and Fabry Disease
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Other Study IDs: Fabry2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Fabry disease is a rare X-linked lysosomal storage disorder. The mutations result in a deficiency of the lysosomal enzyme α-galactosidase causing accumulation of glycosphingolipids in the vascular endothelial cells and many other tissues. An early sign of the disease is painful small fibre neuropathy presenting in two forms: 1. a constant burning sensation in the hand and feet and 2. Fabry crises consisting of attacks of excruciating pain. Given the X-linked inheritance, male patients are severely affected. Recently attention has been drawn to female patients whether they also show signs of nerve involvement.

The purpose of this study is to evaluate the small fibre neuropathy in female Fabry patients. Correlation with X-chromosome inactivation will be attempted. Recombinant human α-galactosidase A is now available for patients. A part of this study is evaluation the long term efficacy of enzyme replacement therapy in female patients with Fabry disease and neuropathy.

Male family members with Fabry disease will be examined.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with confirmed Fabry disease

Exclusion Criteria:

* Patients who cannot cooperate
* Patients who are unable to understand the purpose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-01; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anette T Moller, MD, Principal Investigator — Danish Pain Research Center; Troels S Jensen, MD, PhD, Study Chair — Danish Pain Research Center
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark